CLINICAL TRIAL: NCT01985282
Title: Evaluate the Feasibility of the NLA Tool, a Combined Assessment of Nutritional and Physical Functional Status, to Provide Personalized Advice for the Independence and Mobility of Elderly.
Brief Title: Feasibility Clinical Study of NLA Tool
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 12.33.NRC
Record Dates: First submitted 2013-04-22; First posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Healthy Elder People

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Nutrition Status and Physical Function: Nutrition questionnaire will be administered Physical functional status will be tested
  Interventions: Behavioral: Nutrition Status Questionnaires and Physicial Function Test

INTERVENTIONS:
Behavioral: Nutrition Status Questionnaires and Physicial Function Test — Nutrition status questionnaires will be administered, Physical functional status will be tested

SUMMARY:
The study is to evaluate the feasibility of the NLA tool, a combined assessment of nutritional and physical functional status, to provide personalized advice for the independence and mobility of elderly.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 65 and 90 years,
2. able to walk with or without walking aid,
3. having obtained the subject's written informed consent
4. free of cognitive impairment,

Exclusion Criteria:

1. restricted by a doctor to exercise.
2. unable to carry out performance tests and questionnaires correctly,
3. lower or upper extremity surgery or fracture in the last 3 months
4. having history of neurological disease (e.g., Parkinson disease, stroke) with residual impairment

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Free-living or institutionalized elderly (65-90years)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
NLA Feasibility | Day 1 of Study
  Determining the proportion of elderly subjects (by statistical approach) who, according to the NLA result, would qualify for a personalized program to improve their nutritional and physical status
The Segmentation of Target Population | Day 1 of Study
  Determining the segmentation (defined by cut-off criteria) of these elderly subjects stratified into 3 NLA subgroups according to strength (By measuring upper and lower extremity strength) and endurance performance (By measuring 6 minutes walking distantce) (33% +/- 10% of target group)

CONTACTS AND LOCATIONS:
Overall Officials: Kiyoji Tanaka, PhD, Principal Investigator — Graduate School of Comprehensive Human Sciences, Tsukuba University
Locations (1):
- Graduate School of Comprehensive Human Sciences, Tsukuba University, Tsukuba, Ibaraki, Japan